CLINICAL TRIAL: NCT05227079
Title: Comparison of the Histological Quality of Endoscopic Biopsy Samples Obtained With Novel Multiple-bite Forceps Versus Conventional Double Bite Forceps
Brief Title: Assessing the Histological Quality of Biopsy Samples Obtained With Multibite Forceps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lawrence Charles Hookey (Other)
Responsible Party: Sponsor-Investigator, Lawrence Charles Hookey, Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: DMED-2634-21
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Helicobacter Pylori Infection; Celiac Disease
Keywords: Biopsy; Histological quality; Endoscopy; Forceps
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two groups (group A and group B). Group A will include patients who will have their biopsies taken with the conventional double bite forceps during endoscopy. Group B will include patients who will have their biopsies taken with the multiple bite forceps.
  Each patient in both groups will have the same number of biopsies taken from the same anatomical areas; the only difference will be the number of biopsies that are taken consecutively.
Who Masked: Participant, Investigator
Masking Description: The participant will be blinded as to which forceps (ie. conventional double bite or multiple bite forceps) are used for sampling during endoscopy.
  The pathologists assessing the histological quality of biopsy specimens will also be blinded to which forceps were used to obtain the samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (double bite forceps) (Active Comparator): Participants in group A will proceed to have their biopsies during endoscopy taken with the conventional double bite forceps. Meaning, they will have two biopsies taken each time the forcep is passed through the endoscope. To obtain a total of six biopsies, the forceps will be passed through the endoscope a total of three times.
  Interventions: Device: Conventional double bite forcep
- Group B (multiple bite forceps) (Experimental): Participants in group B will have their biopsies during endoscopy retrieved with the multiple bite forceps. Meaning, they will have six consecutive biopsies taken with each pass through the endoscope.
  Interventions: Device: MultCROC multibite forcep

INTERVENTIONS:
Device: MultCROC multibite forcep — Alligator style 2.4 mm diameter jaws that can hold up to six samples in one pass through endoscope.
  Arms: Group B (multiple bite forceps)
Device: Conventional double bite forcep — Use of conventional double bite forceps that can store up to two specimens in one pass through endoscope
  Arms: Group A (double bite forceps)

SUMMARY:
Biopsies are routinely taken during endoscopy and colonoscopy in order to facilitate histological analysis of various disease processes. The current practice of obtaining biopsies involves taking a maximum of two biopsies at a single time (ie. with a single pass). When investigating certain diseases, such as celiac disease, there is a need to obtain several biopsies (sometimes greater than 6) and the current practice of taking one to two biopsies at a time can lengthen endoscopy time. This study investigates a new approved multiple bite forceps that has the ability to retrieve six biopsies during a single pass which could reduce endoscopy time and improve diagnostic yield. This study will assess the histological quality of multiple biopsies when taken with the multiple bite forceps compared to the standard double bite forceps. This multiple bite forcep is approved for clinical use in Canada.

DETAILED DESCRIPTION:
This will be a prospective randomized noninferiority study that will take place at Hotel Dieu Hospital. Based on a statistical power calculation, a total of 100 patients are required for enrollment. Enrollment will take place at the outpatient endoscopy suite at Hotel Dieu Hospital. Patients will be reviewed for eligibility as per the inclusion and exclusion criteria and those deemed eligible will consent for participation. Members of the research time will attempt to contact patients two to three weeks prior to their schedule endoscopy for consent. If unable to reach them after two attempts, they will then be consented for their participation during the day of their endoscopy at Hotel Dieu Hospital. Once enrolled in the study, each patient will be randomly allocated to one of two groups (group A and group B) using a computer randomizer generator. The aim is to have equal numbers in both groups (ie. 50 patients in each group). Participants in group A will have their biopsies during endoscopy taken with the conventional double bite forceps. On the other hand, participants in group B will have their biopsies taken with the multiple bite forceps. Each patient in both groups will have at least six biopsies taken. In both groups, biopsies will be taken for assessment of H. pylori and/or celiac disease. Patients recruited will be those who would require these biopsies to be taken regardless of this study. The samples will be sent to pathology where two independent expert gastrointestinal pathologists will examine the slides and grade each specimen using a five-point scale. The overall histological score given to samples will then be assessed to compare those retrieved with the multiple bite forceps and conventional forceps.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were referred for outpatient upper endoscopy at Hotel Dieu Hospital requiring biopsies to investigate for celiac disease or H. Pylori infection.

Exclusion Criteria:

* Patients with clinical or endoscopic evidence of gastric mucosal atrophy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Histological quality | Duration of endoscopy and pathological assessment of specimens
  Comparison of the histological quality of specimens retrieved with multiple bite forceps compared to double bite forceps

SECONDARY OUTCOMES:
Time duration | Duration of endoscopy
  Total time taken to retrieve six biopsies with the multiple bite forceps compared to time taken to retrieve six biopsies using double bite forceps

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C Hookey, MD, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lebwohl B, Kapel RC, Neugut AI, Green PH, Genta RM. Adherence to biopsy guidelines increases celiac disease diagnosis. Gastrointest Endosc. 2011 Jul;74(1):103-9. doi: 10.1016/j.gie.2011.03.1236. Epub 2011 May 20. PMID 21601201
- [Background] Rostom A, Murray JA, Kagnoff MF. American Gastroenterological Association (AGA) Institute technical review on the diagnosis and management of celiac disease. Gastroenterology. 2006 Dec;131(6):1981-2002. doi: 10.1053/j.gastro.2006.10.004. No abstract available. PMID 17087937
- [Background] Rubio-Tapia A, Hill ID, Kelly CP, Calderwood AH, Murray JA; American College of Gastroenterology. ACG clinical guidelines: diagnosis and management of celiac disease. Am J Gastroenterol. 2013 May;108(5):656-76; quiz 677. doi: 10.1038/ajg.2013.79. Epub 2013 Apr 23. PMID 23609613
- [Background] Zaidman JS, Frederick WG, Furth EE, Su CG, Ginsberg GG. Comparison of Pelican single-use multibite biopsy forceps and traditional double-bite forceps: evaluation in a porcine model. Gastrointest Endosc. 2006 Oct;64(4):582-8. doi: 10.1016/j.gie.2006.06.060. PMID 16996354
- [Result] Fantin AC, Neuweiler J, Binek JS, Suter WR, Meyenberger C. Diagnostic quality of biopsy specimens: comparison between a conventional biopsy forceps and multibite forceps. Gastrointest Endosc. 2001 Nov;54(5):600-4. doi: 10.1067/mge.2001.118945. PMID 11677476